CLINICAL TRIAL: NCT04021940
Title: A Randomized Comparison of Dose Adjusted vs. Fixed Dose Unilateral Laparoscopic Ovarian Drilling in Polycystic Ovary Syndrome Patients
Brief Title: Dose Adjusted vs. Fixed Dose Unilateral Laparoscopic Ovarian Drilling in PCOS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.19.05.615
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose adjusted ULOD (Experimental): dose adjusted ULOD using 60J/cm3 applied to the larger ovary. The number of punctures (Np) per ovary will be calculated according to the following formula: Np = 60 J/cm3 divided by 30 W x 4 s.
  Interventions: Procedure: ULOD
- Fixed dose ULOD (Active Comparator): 600 J for the larger ovary will be delivered through four punctures, each for 4 s and 40 W
  Interventions: Procedure: ULOD

INTERVENTIONS:
Procedure: ULOD — ULOD

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder and a leading cause of infertility in women of reproductive age affecting up to 20% of them. Laparoscopic ovarian drilling (LOD) is considered a second-line treatment of infertile patients with clomiphene citrate-resistant (CCR) PCOS i.e. those who did not ovulate in response to CC doses of up to 150 mg for at least three consecutive cycles. The advantage of LOD is the induction of unifollicular ovulation without the risk of ovarian hyperstimulation syndrome or high-order multiple pregnancies.

The common practice of LOD was to drill both ovaries i.e. bilateral (BLOD) with a fixed dose of 600 Joules per each ovary (1200 Joules in both) delivered through four punctures, each for 4 s and using 40 W. However, its main adverse effect is diminished ovary reserve due to tissue damage (2). In 1994, Balen and Jacobs reported the effectiveness of fixed-dose unilateral LOD (ULOD) in the management of those women. Subsequently, several randomized trials demonstrated its efficacy with comparable ovulation and pregnancy rates to BLOD.

Recently, a new concept called"dose-adjusted" ULOD was proposed. It means to tailor the energy applied to one ovary, according to its preoperative volume using 60 J/ cm3. When compared with the fixed-dose BLOD among 96 infertile women with CCR- PCOS, a significantly higher ovulation rate during the first postoperative menstrual cycle was in favor of the ULOD group (73 vs. 49%). Meanwhile, a comparable ovulation rate over the 6-month period was found (82 vs. 64%) (6). In addition, both groups experienced a reduction in serum anti-mullerian hormone (AMH) level after LOD which was significantly more in the BLOD group in the first and the 6-month follow-up periods. However, another RCT (n=108 CCR- PCOS patients) reported a comparable ovulation and pregnancy rates at 3-month follow-up period (65.4 vs. 77.3% and 15.4 vs. 26.4%, in ULOD and BLOD respectively) with a reduction in the effectiveness of dose-adjusted ULOD after 6 months. A highly significant difference between ULOD and BLOD groups with regard to the AMH level at 3- and 6-month was also reported. Thereby, the efficacy of dose-adjusted ULOD in improving fertility outcomes in infertile women with CCR- PCOS as well as its effect on ovarian reserve warrants more investigation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS will be based on the revised 2003 consensus on diagnostic criteria and long-term health risks related to PCOS and its modification (ESHRE, 2018).
* CCR will be considered if persistent anovulation with 150 mg CC daily for 5 days per cycle, for at least three cycles.
* Only patients with a phenotype characterized by oligomenorrhoea/anovulation, hyperandrogenaemia and polycystic ovaries on ultrasound examination (PCOM) and a phenotype characterized by oligomenorrhoea/anovulation and PCOM will be enrolled in the study.
* Age: 20-34 years.
* Body mass index < 30 kg/m2
* Patent fallopian tubes by hysterosalpingography.
* Normal semen analysis of husbands.

Exclusion Criteria:

* Age ≥ 35 years.
* BMI ≥ 30
* Previous history of LOD
* PCOS phenotypes with regular menses or without PCOM ovaries on USS.
* Other causes of infertility
* Women with adrenal hyperplasia, thyroid disease, Cushing's syndrome, hyperprolactinemia and a tumor-related excess of androgen.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-08-05 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
ovulation rate | At 6 months postoperative
  serum progesterone level >5 ng/mL on D 21 of the cycle

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. FRCOG. PhD, Study Chair — Faculty of Medicine, Mansoura University; Eman Lotfy, MBBCh, Principal Investigator — New Mansoura General Hospital

REFERENCES:
- [Background] Abu Hashim H, Foda O, El Rakhawy M. Unilateral or bilateral laparoscopic ovarian drilling in polycystic ovary syndrome: a meta-analysis of randomized trials. Arch Gynecol Obstet. 2018 Apr;297(4):859-870. doi: 10.1007/s00404-018-4680-1. Epub 2018 Jan 27. PMID 29374790